CLINICAL TRIAL: NCT04753437
Title: A Phase 1, Double-Blind, Parallel Group Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Quadruple Therapy (Bismuth, Clarithromycin, and Amoxicillin) With Vonoprazan Versus Quadruple Therapy With Esomeprazole
Brief Title: A Study of Vonoprazan in Adults With Helicobacter Pylori
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Vonoprazan-1001; U1111-1257-0258 (Registry Identifier: WHO)
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori
Keywords: Drug Therapy
MeSH Terms: interventions — Clarithromycin; Amoxicillin; Esomeprazole; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clarithromycin + Amoxicillin + Bismuth + Vonoprazan (Experimental): Clarithromycin 500 milligram (mg), tablets, orally, BID, along with amoxicillin 1000 mg, capsules, orally, BID, bismuth potassium citrate 600 mg, capsules, orally, BID, and vonoprazan 20 mg, tablets, orally, BID on Days 1 to 14.
  Interventions: Drug: Clarithromycin; Drug: Amoxicillin; Drug: Bismuth potassium citrate; Drug: Vonoprazan
- Clarithromycin + Amoxicillin + Bismuth + Esomeprazole (Active Comparator): Clarithromycin 500 mg, tablets, orally, BID, along with amoxicillin 1000 mg, capsules, orally, BID, bismuth potassium citrate 600 mg, capsules, orally, BID, and esomeprazole 20 mg, tablets, orally, BID on Days 1 to 14.
  Interventions: Drug: Clarithromycin; Drug: Amoxicillin; Drug: Bismuth potassium citrate; Drug: Esomeprazole

INTERVENTIONS:
Drug: Clarithromycin — Clarithromycin tablets.
Drug: Amoxicillin — Amoxicillin capsules.
Drug: Bismuth potassium citrate — Bismuth potassium citrate tablets.
Drug: Esomeprazole — Esomeprazole tablets.
  Arms: Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
Drug: Vonoprazan — Vonoprazan tablets.
  Other Names: TAK-438
  Arms: Clarithromycin + Amoxicillin + Bismuth + Vonoprazan

SUMMARY:
Helicobacter Pylori (H Pylori) is a bug found in the digestive system. It can cause soreness and redness in the stomach (gastritis). It can also cause ulcers in the stomach and other parts of the digestive system. Vonoprazan is a medicine to treat people with H Pylori. It is taken together with other medicines to fight infections caused by H Pylori.

The main aim of this study is to learn if vonoprazan changes how the other medicines are processed by the body. It will be compared with another medicine called esomeprazole. Other aims are to check for side effects from the study medicines.

At the first visit, the study doctor will check who can take part. Participants who take part will be picked for 1 of 2 treatments by chance.

* Vonoprazan taken with bismuth, clarithromycin, and amoxicillin
* Esomeprazole taken with bismuth, clarithromycin, and amoxicillin

Both treatments will last for 14 days. Participants will stay in the clinic throughout their treatment.

After treatment, the clinic staff will telephone the participants 2 days later for a check-up. The participants will visit the clinic 4 weeks later for a final check-up.

DETAILED DESCRIPTION:
This is a study in healthy participants with Helicobacter pylori (HP positive) to evaluate the safety, tolerability and PK of a quadruple therapy with bismuth, clarithromycin, amoxicillin, and vonoprazan versus quadruple therapy with bismuth, clarithromycin, amoxicillin, and esomeprazole.

The treatment phase consists of quadruple therapy twice daily (BID) with bismuth potassium citrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and vonoprazan (20 mg) (Group B) or quadruple therapy BID with bismuth potassium citrate (600 mg), clarithromycin (500 mg), amoxicillin (1000 mg), and esomeprazole (20 mg) (Group A) from Days 1 to 14. Participants will be discharged on Day 15 after all procedures have been performed.

This single-center will be conducted in China. Participants will remain confined to the study site from check-in (Day -1) through Day 15 and will followed up through call on Day 17 and return on Day 42 for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. HP positive participants.
2. Weighs at least 50 kilogram (kg) and has a body mass index between greater than (>) 18 and less than equal to (<=) 30 kilogram per square meter (kg/m^2), inclusive, at screening and Day -1 (check-in).
3. Is willing to abstain from strenuous exercise from 72 hours before first dose (Day 1) until the Follow-up call on Day 17.

Exclusion Criteria:

1. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
2. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular consumption of 21 units or more units per week) at any time prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study (up to Day 17).
3. Has history of gastroesophageal reflux disease (GERD), symptomatic GERD, erosive esophagitis, duodenal ulcer, gastric ulcer, Barrett's esophagus, or Zollinger-Ellison syndrome, or has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs.
4. Has undergone therapeutic upper gastrointestinal endoscopic therapy (example, endoscopic hemostasis or excision including biopsy) within 30 days prior to Screening.
5. Has undergone major surgical procedures within the past 1 month or are scheduled to undergo surgical procedures that may affect gastric acid secretion (example, abdominal surgery, vagotomy, or craniotomy).
6. Has a history of cancer, except basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin that has been in remission for at least 5 years prior to Day 1.
7. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen at Screening.
8. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 6 weeks prior to Check-in. Cotinine test is positive at Screening or Check-in.
9. Has poor peripheral venous access.
10. Has donated or lost 450 milliliter (mL) or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 90 days prior to Day 1.
11. Has abnormal Screening or Check-in laboratory values that suggest a clinically significant underlying disease or subject with the following laboratory abnormalities: alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin > the upper limit of normal (ULN).
12. Has reduced renal function assessed by having an estimated glomerular filtration rate <90 milliliter per min per 1.73 square meter (mL/min/1.73 m^2) (as estimated by Chronic Kidney Disease-Epidemology Collaboration) at Screening or Check-in.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- West China Hospital, Sichuan University, Phase I Unit, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/6036adec20847c001e116be1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in China from 06 April 2021 to 05 November 2021.
Pre-assignment Details: Helicobacter pylori (H pylori) positive participants were enrolled and randomized to one of the two treatment groups to either receive quadruple therapy with bismuth, clarithromycin, amoxicillin, and vonoprazan versus quadruple therapy with bismuth, clarithromycin, amoxicillin, and esomeprazole.
Groups:
- Clarithromycin + Amoxicillin + Bismuth + Vonoprazan: Clarithromycin 500 milligram (mg), tablets, orally, twice daily (BID), along with amoxicillin 1000 mg, capsules, orally, BID, bismuth potassium citrate 600 mg, capsules, orally, BID, and vonoprazan 20 mg, tablets, orally, BID on Days 1 to 14.
Period: Overall Study
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
Started | 22 | 22
Completed | 20 | 17
Not Completed | 2 | 5
Not completed — Pretreatment Event/Adverse Event | 0 | 1
Not completed — Liver Function Test Abnormalities | 2 | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Clarithromycin + Amoxicillin + Bismuth + Vonoprazan: Clarithromycin 500 mg, tablets, orally, BID, along with amoxicillin 1000 mg, capsules, orally, BID, bismuth potassium citrate 600 mg, capsules, orally, BID, and vonoprazan 20 mg, tablets, orally, BID on Days 1 to 14.
- Total: Total of all reporting groups
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.60) | 31.6 (9.59) | 33.1 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 22 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 22 | 22 | 44
Height [Mean (Standard Deviation); unit: cm] | 167.2 (6.58) | 165.6 (7.17) | 166.4 (6.85)
Weight [Mean (Standard Deviation); unit: kg] | 62.8 (9.23) | 63.2 (8.23) | 63.0 (8.64)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI= weight (kg)/[height (m)^2]
  kg/m^2 | 22.4 (2.07) | 23.1 (3.09) | 22.7 (2.63)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Bismuth
Time Frame: Day 14: 0 to 12 hours after the morning dose
Population: Pharmacokinetic (PK) Analysis Set included participants who received the study drug (bismuth, vonoprazan or esomeprazole, clarithromycin, amoxicillin) and had at least 1 measurable plasma drug concentration after start of dosing without protocol violations or events with potential to affect the PK concentrations and who had completed minimum protocol procedures.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
Number analyzed (Participants) | 20 | 18
nanogram per milliliter (ng/mL) | 42.8 [32.6 to 56.2] | 32.9 [24.7 to 43.8]
Statistical Analysis 1: Comparison: Clarithromycin + Amoxicillin + Bismuth + Vonoprazan vs Clarithromycin + Amoxicillin + Bismuth + Esomeprazole; Test type: Equivalence — Results were based on analysis of variance model with treatment as a fixed effect; Geometric Least Squares (LS) Mean Ratio = 1.30, 90% CI 2-sided [0.94 to 1.81]

2. Primary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve During a Dosing Interval τ for Bismuth
Time Frame: Day 14: 0 to 12 hours after the morning dose
Population: PK Analysis set included participants who received the study drug (bismuth, vonoprazan or esomeprazole, clarithromycin, amoxicillin) and had at least 1 measurable plasma drug concentration after start of dosing without protocol violations or events with potential to affect the PK concentrations and who had completed minimum protocol procedures.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
Number analyzed (Participants) | 20 | 18
hour*nanogram/milliliter (h*ng/mL) | 146 [117 to 183] | 137 [108 to 173]
Statistical Analysis 1: Comparison: Clarithromycin + Amoxicillin + Bismuth + Vonoprazan vs Clarithromycin + Amoxicillin + Bismuth + Esomeprazole; Test type: Equivalence — Results were based on analysis of variance model with treatment as a fixed effect; Geometric LS Mean Ratio = 1.07, 90% CI 2-sided [0.82 to 1.40]

3. Primary Outcome: Aeτ: Total Amount of Bismuth Excreted in Urine During a Dosing Interval τ for Bismuth
Time Frame: Day 14: 0 to 12 hours after the morning dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrograms (μg)
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
Number analyzed (Participants) | 20 | 18
micrograms (μg) | 1026 (546.0) | 1037 (562.5)

4. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: From the first dose of study drug up to Day 17
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
Number analyzed (Participants) | 22 | 22
percentage of participants | 95.5 | 95.5

5. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug Due to a Treatment-Emergent Adverse Event (TEAE)
Time Frame: From the first dose of study drug up to Day 17
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
Number analyzed (Participants) | 22 | 22
percentage of participants | 9.1 | 22.7

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to Day 17
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any adverse event spontaneously reported by the participant or in response to an open question from study personnel or revealed by observation, physical examination, or other diagnostic procedures was recorded, irrespective of the causality with study drug. Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 21/22 | 21/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clarithromycin + Amoxicillin + Bismuth + Vonoprazan (N=22) | Clarithromycin + Amoxicillin + Bismuth + Esomeprazole (N=22)
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Alanine aminotransferase increased (Investigations) | 9 | 8
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 1 | 3
Amylase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 9 | 7
Blood lactate dehydrogenase increased (Investigations) | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 15 | 18
Faeces discoloured (Gastrointestinal disorders) | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Hunger (General disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Thirst (General disorders) | 2 | 0
Tonsillitis (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04753437/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT04753437/SAP_001.pdf